CLINICAL TRIAL: NCT02479308
Title: The Effect of ALKS 5461 on QT Intervals in Healthy Volunteers
Brief Title: A Study to Evaluate the Effect of ALKS 5461 on QT Intervals in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALK5461-213
Record Dates: First submitted 2015-06-05; First posted 2015-06-24 (Estimated); Last update posted 2015-11-23 (Estimated); Status verified 2015-11

CONDITIONS: Healthy
Keywords: Alkermes; Samidorphan; ALKS 5461; QT/QTc; Buprenorphine; Pharmacodynamics
MeSH Terms: interventions — Moxifloxacin; ALKS 5461

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Moxifloxacin (Active Comparator): Oral tablet
  Interventions: Drug: Moxifloxacin
- ALKS 5461 (Experimental): Sublingual tablet
  Interventions: Drug: ALKS 5461
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Moxifloxacin — Single administration
  Arms: Moxifloxacin
Drug: ALKS 5461 — Daily administration for a total of 12 dosing days
  Arms: ALKS 5461
Drug: Placebo — Placebo will be matched to Moxifloxacin or ALKS 5461
  Arms: Placebo

SUMMARY:
This study will evaluate the effects of ALKS 5461 on QT intervals in healthy volunteers as well as evaluate the safety and tolerability of ALKS 5461.

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index (BMI) of 18.0-30.0 kg/m2 at screening
* Is physically healthy
* Agree to abide by the contraception requirements for the duration of the study
* Additional criteria may apply

Exclusion Criteria:

* Have a positive pregnancy test and/or be currently breastfeeding
* Have a history of or current infection with Hepatitis B virus, Hepatitis C virus, or human immunodeficiency virus (HIV)
* Have current evidence of or history of any clinically significant medical or psychiatric condition or observed abnormality
* Have any skin condition likely to interfere with ECG electrode placement or adhesion
* Have current abuse or dependence (within the past 5 years) on any drugs (exclusive of nicotine or caffeine)
* Have used any prescription or over-the-counter (OTC) medication, including natural health products or dietary supplements (with the exception of prescription contraceptives or hormonal replacements, acetaminophen, ibuprofen, or multivitamins), or have consumed grapefruit or any grapefruit products within 14 days prior to the first study drug dose
* Have consumed alcohol-, caffeine-, or xanthine-containing products within 24 hours prior to the first study drug dose
* Have used nicotine within 90 days prior to the first study drug dose
* Have used opioids 30 days prior to screening, or have an anticipated need for opioid medication during the study
* Additional criteria may apply

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 129 (Actual)
Dates: Start 2015-06; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change in QT interval corrected for heart rate using the Fridericia formula (QTcF) | Up to 14 days

SECONDARY OUTCOMES:
Change in heart rate | Up to 14 days
Incidence of abnormal ECG | Up to 13 days
Tabulation of ECG morphology | Up to 14 days
  Findings not present at baseline
Correlation of plasma drug levels with QT interval | Up to 14 days
Maximum observed plasma concentration (Cmax) for ALKS 5461 | Up to 14 days
Incidence of adverse events (AEs) | Up to 14 weeks
Change in PR interval | Up to 14 days
Change in QRS interval | Up to 14 days
Time to reach the maximum plasma concentration (Tmax) for ALKS 5461 | Up to 14 days
AUC(0-last): Area under the plasma concentration-time curve from time 0 to the time of the last quantifiable concentration for ALKS 5461 | Up to 14 days
AUC(0-inf): Area under the plasma concentration-time curve from time 0 to infinity for ALKS 5461 | Up to 14 days
Terminal elimination half-life (T1/2) for ALKS 5461 | Up to 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Sanjeev Pathak, MD, Study Director — Alkermes, Inc.; Arielle Stanford, MD, Study Director — Alkermes, Inc.
Locations (1):
- Alkermes Investigational Site, Overland Park, Kansas, United States